CLINICAL TRIAL: NCT05567705
Title: The Attitudes of Doctors Working in the Surgical Clinic of a University Hospital for Patient Blood Management: a Survey-based Study
Brief Title: The Attitudes of Doctors Working in the Surgical Clinic of Patient Blood Management
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2019/18
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-10

CONDITIONS: A Survey-based Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: The attitudes of doctors working in the surgical clinic of a university hospital for patient blood management: a survey-based study — No intervention required

SUMMARY:
The attitudes of doctors working in the surgical clinic of a university hospital for patient blood management: a survey-based study

ELIGIBILITY:
Inclusion Criteria:

- Being a doctor working in the surgical clinics of the university hospital

Exclusion Criteria:

* INQUIRING SURVEY QUESTIONS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both genders will be included in the study
Study Population: Being a doctor working in the surgical clinics of the university hospital
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The attitudes of doctors working in the surgical clinic of a university hospital for patient blood management: a survey-based study | about 2 months
  The approach of physicians working in surgical clinics to patient blood management

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No